CLINICAL TRIAL: NCT00982098
Title: Prevention of Urinary Incontinence After Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Carlo Cisari, AUO "Maggiore della Carità"
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NO08974
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Urinary Incontinence
Keywords: Prostatectomy; Prostatic cancer; Urinary incontinence; Exercise; Electric stimulation therapy; Counseling
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms; Motor Activity | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Early Rehabilitation (Experimental): Before surgery: 15 minutes pelvic floor muscle training and 15 minutes biofeedback, for 4 sessions.
  After surgery: physical therapist's assisted pelvic floor muscle biofeedback (15 min/day for 10 days), followed by patient's instruction for pelvic floor muscle training and home based exercised pelvic floor muscle for 10 days. Then pelvic floor muscle biofeedback (15 min/day for 10 days) and functional electrical stimulation of pelvic floor (30 min/day for 10 days).
  Patients will be instructed to carry on exercises at home for the following 11 months.
  Interventions: Procedure: BioFeedback; Functional Electrical Stimulation; Pelvic Floor Muscle training exercises
- Counseling and home-based exercises (No Intervention): Before surgery: 15 minutes pelvic floor muscle training and 15 minutes biofeedback, for 4 sessions.
  After surgery: Patients will be instructed to carry on pelvic floor exercises at home for the year after prostatectomy.

INTERVENTIONS:
Procedure: BioFeedback; Functional Electrical Stimulation; Pelvic Floor Muscle training exercises — After surgery: physical therapist's assisted pelvic floor muscle biofeedback (15 min/day for 10 days), followed by patient's instruction for pelvic floor muscle training and home based exercised pelvic floor muscle for 10 days. Then pelvic floor muscle biofeedback (15 min/day for 10 days) and functional electrical stimulation of pelvic floor (30 min/day for 10 days).
  Arms: Early Rehabilitation

SUMMARY:
Urinary incontinence is a frequent complication after radical prostatectomy. Rehabilitative treatments are frequently utilized to reduce incontinence. However, their efficacy has not been completely investigated. In this study the investigators will compare the effect of an early rehabilitation programme (instruction of the patient, pelvic floor muscle training, electrical stimulation and biofeedback) versus instruction of the patient only.

The investigators hypothesis is that early rehabilitation programme is more effective than patient's instruction alone in preventing urinary incontinence after radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* men who will undergo radical prostatectomy for prostatic cancer

Exclusion Criteria:

* previous urinary and/or faecal incontinence
* neurologic bladder
* previous pelvic surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Complete continence (PAD test 24 hours <10 cc) | 12 months

SECONDARY OUTCOMES:
PAD test 24 hours | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Cisari, prof., Study Director — AUO "Maggiore della Carità" - Novara; Carlo Terrone, prof., Study Chair — AUO "Maggiore della Carità" - Novara
Locations (1):
- SC Medicina Fisica e Riabilitativa AUO "Maggiore della Carità", Novara, Italy